CLINICAL TRIAL: NCT03202745
Title: The Effect of Informative Letters on the Prescription and Receipt of Opioids
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Intervention never conducted
Sponsor: Abdul Latif Jameel Poverty Action Lab (Other)
Collaborators: Centers for Medicare and Medicaid Services (U.S. Federal Agency); General Services Administration (GSA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: JPAL-LETTERS-OPIOIDS
Record Dates: First submitted 2017-06-27; First posted 2017-06-29 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Economics; Fraud; Delivery of Health Care; Health Expenditures; Prescribing; Centers for Medicare and Medicaid Services (U.S.)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): The control arm will not receive any communications as a result of this study.
- Patient Consequences (Experimental): The patient consequences arm prescribers receive an initial patient consequences letter followed by 2 followup letters at approximately 3 month intervals. The letters focus on the consequences of inappropriate prescribing for patients.
  Interventions: Other: Patient Consequences Letter
- Prescriber Consequences (Experimental): The prescriber consequences arm prescribers receive an initial prescriber consequences letter followed by 2 followup letters at approximately 3 month intervals. The letters focus on the consequences of inappropriate prescribing for prescribers.
  Interventions: Other: Prescriber Consequences Letter

INTERVENTIONS:
Other: Patient Consequences Letter — This letter focuses on the consequences of inappropriate prescribing for patients. It also includes a peer comparison.
  Arms: Patient Consequences
Other: Prescriber Consequences Letter — This letter focuses on the consequences of inappropriate prescribing for prescribers. It also includes a peer comparison.
  Arms: Prescriber Consequences

SUMMARY:
Inappropriate prescribing exposes patients to health risks and results in wasteful public expenditures. This study will evaluate an approach to fighting abusive prescription: sending letters to suspected potentially inappropriate prescribers warning them that they are outliers compared to their peers and have been flagged for review. The study will target high prescribers of opioids in the Schedule II controlled substances class. Two types of letters will be tested: one focusing on the health consequences of inappropriate prescribing for patients, and the other focusing on the consequences for prescribers including e.g. potential administrative actions. Using claims data, the investigators will assess the effect of the letters on prescribing of opioids, receipt of opioids by patients, substitution behavior by prescribers and patients, and health outcomes of patients.

ELIGIBILITY:
Inclusion Criteria:

* Outlier with respect to prescribing of Schedule II opioids relative to peers, measured in prescription drug events (PDE), in 2014Q3-2015Q2 and 2015Q3-2016Q2
* Outlier with respect to prescribing of Schedule II opioids relative to peers, measured in 30-day equivalents, in 2014Q3-2015Q2 and 2015Q3-2016Q2

Exclusion Criteria:

* Deceased
* Fewer than 75 Schedule II Opioid PDE in 2015Q3-2016Q2
* Specialty listed as "Student in an Organized Health Care Education/Training Program"

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2018-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Morphine Milligrams Equivalent (MME) | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Adam Sacarny, PhD, Principal Investigator — Columbia University

IPD SHARING:
Plan to Share IPD: Undecided